CLINICAL TRIAL: NCT03527615
Title: Clinical Pharmacist Led Hospital-Wide Direct Oral Anticoagulant Stewardship Program
Brief Title: Clinical Pharmacist Anticoagulant Stewardship
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: DOACPHARM-HMO-CTIL
Record Dates: First submitted 2018-04-16; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Safety Issues; Anticoagulant Toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical Pharmacist Medication Review — Programmatic review of physician orders for direct anticoagulants by clinical pharmacists.

SUMMARY:
Initiative to improve direct anticoagulant utilization involving programmatic review by clinical pharmacists in collaboration with multidisciplinary team.

DETAILED DESCRIPTION:
The Hadassah Hebrew University Medical Centers' Clinical Pharmacy team initiated a hospital-wide program, in collaboration with the institutions' coagulation specialists, including two hematologists and a clinical pharmacologist, for monitoring and promoting safe and effective prescription of direct oral anticoagulants (DOAC) during hospitalization. Electronic medical records throughout the hospital are screened for DOAC orders. All DOAC orders are assessed by a clinical pharmacist for potentially-inappropriate prescribing. When potentially-inappropriate prescribing or a drug-related problem is identified, the clinical pharmacist provided consultation on management options. In specific cases, additional guidance is provided by coagulation specialists. Consultations are recorded in the electronic medical record. Performance measures are collected and summarized.

ELIGIBILITY:
Inclusion Criteria:

Patients hospitalized in Hadassah Medical Center with a physician's order for direct oral anticoagulants (apixaban, rivaroxaban, or dabigatran).

Exclusion Criteria:

Patients hospitalized in departments without computerized physician order entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in Hadassah Medical Center with a physician's order for direct oral anticoagulants.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Percent of clinical pharmacist consultations accepted by attending physician. | At forty-eight months
  Calculated by dividing the number of clinical pharmacist consultations accepted, by the number of clinical pharmacist consultations given, during the period. Data for consultation counts will be obtained from patient electronic medical record.

SECONDARY OUTCOMES:
Percent of clinical pharmacist consultations accepted by attending physician. | At six months
  Calculated by dividing the number of clinical pharmacist consultations accepted, by the number of clinical pharmacist consultations given, during the period. Data for consultation counts will be obtained from patient electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Muszkat, MD, Principal Investigator — Hadassah University Medical Center
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perlman A, Horwitz E, Hirsh-Raccah B, Aldouby-Bier G, Fisher Negev T, Hochberg-Klein S, Kalish Y, Muszkat M. Clinical pharmacist led hospital-wide direct oral anticoagulant stewardship program. Isr J Health Policy Res. 2019 Feb 1;8(1):19. doi: 10.1186/s13584-019-0285-9. PMID 30709417